CLINICAL TRIAL: NCT00155584
Title: Topical 5-Aminolevulinic Acid Photodynamic Therapy for the Treatment of Verruca Vulgaris: Comparison of Red and Green Light-Emitting Diode Array
Brief Title: Topical 5-ALA Photodynamic Therapy for the Treatment of Verruca Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 28MD01
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 1994-12

CONDITIONS: Warts
Keywords: warts; photodynamic therapy; 5-ALA
MeSH Terms: conditions — Warts

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
Photodynamic therapy (PDT) has been developed as a promising new cancer treatment modality, which involves the uptakes of a photosensitizer by tumor cells, followed by the activation of photosensitizer with approximate wavelength of light. The mechanisms of the PDT-induced cytotoxic effect relate to singlet oxygen and other reactive oxygen intermediates generated by PDT, which give rise to cellular stress and cause cell death. Previously, using the homemade LED light source, we have shown that ALA-PDT is effective for the treatment of premalignant lesions such as mucosal dysplasia and carcinoma in situ of oral cavity. Due to the advantages of low cost, high reliability, and portability, LED light source provides an alternative approach for the light irradiation of PDT.

Verruca vulgaris are benign skin papillomas caused by the human papilloma virus (HPV). They are very common and can affect many different sites including the face, hands, feet and genitalia. Although the present therapeutic approaches are more or less effective in eradicating the lesions, relapses are very common. Furthermore, at times the anatomical location and depth of lesions often make the treatment difficult, time-consuming and painful. Therefore, it is necessary to develop new modalities for wart treatment.

The purpose of this clinical trial is to develop topical ALA-PDT as an alternative treatment of wart but without the unwanted side effects of pain and burning. To fulfill this goal, the following works will be performed. First, topical ALA formulation and LED array will be specifically designed and developed for the skin lesions. Second, the efficacy of the ALA formulation designed for wart treatment will be evaluated with in vivo fluorescence imaging system. Third, the therapeutic efficacy of ALA-PDT will be evaluated by using a LED array designed for skin irradiation. Forth, the unwanted side effects of pain and burning will be further compared between red and green LED array.

DETAILED DESCRIPTION:
Verruca vulgaris or warts are benign skin papillomas caused by the human papilloma virus (HPV). They are very common and can affect many different sites including the face, hands, feet and genitalia. Although the present therapeutic approaches are more or less effective in eradicating the lesions, scars and relapses are very common. Furthermore, at times the anatomical location and depth of lesions often make the treatment difficult, time-consuming and painful. Therefore, it is necessary to develop new modalities for wart treatment.

Photodynamic therapy (PDT) has been developed as a promising new cancer treatment modality, which involves the uptakes of a photosensitizer by tumor cells, followed by the activation of photosensitizer with approximate wavelength of light. The endogenous conversion of 5-aminolevulinic acid (ALA) to protoporphyrin IX (PpIX) has broadened the use of PDT. The mechanisms of the PDT-induced cytotoxic effect relate to singlet oxygen and other reactive oxygen intermediates generated by PDT, which give rise to cellular stress and cause cell death. Previously, using the homemade LED light source, we have shown that topical ALA-PDT is effective for the treatment of warts. However, the excruciating pain induced by ALA and red LED could be due to deeper penetration of the ALA formulation or the deeper penetration of red light. Thus the pain might be related to the injured nerve fibers underlying the skin. This study is to provide evidence of these two green or red LED efficacy in removing the warts and also their side-effect of pain.

ELIGIBILITY:
Inclusion Criteria:

Warts -

Exclusion Criteria:

other skin lesions or combined with infection -

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1994-12; Study Completion 1996-12

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, Ph.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan